CLINICAL TRIAL: NCT02260102
Title: Temocillin Pharmacokinetics in Paediatrics
Acronym: TEMOPEDI
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Université Catholique de Louvain (Other)
Responsible Party: Principal Investigator, Paul M. Tulkens, Invited Professor, Université Catholique de Louvain
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: temocillin-pediatrics
Record Dates: First submitted 2014-10-01; First posted 2014-10-09 (Estimated); Last update posted 2022-05-31 (Actual); Status verified 2022-05

CONDITIONS: Infection; Liver Dysfunction; Urinary Tract Infection
MeSH Terms: conditions — Infections; Liver Diseases; Urinary Tract Infections | interventions — temocillin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- urinary tract infections (Active Comparator): Children requiring antibiotic treatment for urinary tract infections. Intervention: blood sampling for assay of temocillin
  Interventions: Drug: Temocillin
- cholangitis (Active Comparator): Cirrhotic children requiring antibiotic treatment due to suspicion of cholangitis.
  Intervention: blood sampling for assay of temocillin
  Interventions: Drug: Temocillin
- hepatic transplant (Active Comparator): Children requiring antibiotic prophylaxis following a hepatic transplant. Intervention: blood sampling for assay of temocillin
  Interventions: Drug: Temocillin

INTERVENTIONS:
Drug: Temocillin — Venous blood will be drawn (as per the protocol) for assay of temocillin on day 1 and day 4 of treatment. This is not part of our standard of care and is, therefore, an intervention. Patients are enrolled only if receiving temocillin as part of their normal standard of care (and the drug will be administered based on current recommendations [no change due to enrollment in the study]).
  Other Names: NEGABAN

SUMMARY:
Temocillin (6-methoxy-ticarcillin) is a beta-lactam antibiotic with exceptional resistance to most beta-lactamases. In this context, it is now increasingly used as carbapenem-sparing antibiotic in patients with suspected infection by Enterobactreriaceae suspected to produce extended-spectrum beta-lactamases. Little is known about dosing and elimination of temocillin in children. While available literature of temocillin use in paediatrics refers mainly to its clinical efficacy in the treatment of urinary tract infections, the drug is also used for the treatment of suspicion of cholangitis in cirrhotic paediatric patients, and as antibiotic prophylaxis following an hepatic transplant in children (both off-label indications). There is, therefore, a pressing need to explore the pharmacokinetics and pharmacodynamics of temocillin in the paediatric population, in order to provide clear guidance on an appropriate dosing regimen. The study objectives are: (1) characterisation of the pharmacokinetics (PK) of temocillin in 3 paediatric populations, (2) proposal and development of a dosing schedule that can ensure therapeutic concentrations (40% ƒT > MIC) and optimize treatment chances of success, and (3) characterization of MICs of microbiological strains (when available) to temocillin.

DETAILED DESCRIPTION:
1. Introduction Temocillin is a beta-lactam antibiotic active against Gram-negative bacteria. Its spectrum covers family members of the Enterobacteriaceae (including many of those producing beta-lactamases), Haemophilus influenzae and Neisseria spp 1,2, but not Pseudomonas. It is currently licensed for use in septicemia, urinary tract infection (UTIs), and lower respiratory tract infection.3 There is also evidence of its clinical efficacy in the treatment of biliary tract infections in adults.4,5 Temocillin biliary levels can be several times-fold superior to serum concentrations in patients with cholelithiasis, although they can also be characterised by high interindividual variation.6,7 In addition, its prolonged half-life (4.5-5 hours) and its Gram-negative spectrum make temocillin particularly suited for the treatment of hepatobiliary infections.5 One study documents the efficacy of temocillin in this indication (16 patients with biliary tract infections; daily dose of 2g of temocillin).7

The interest of this molecule has been greatly enhanced in the recent years due to the increased incidence of infections caused by organisms producing extended-spectrum beta-lactamases (ESBL), making it to become a sparing-drug for carbapenems.8-10 Temocillin presents MICs ranging from 2 to 32 mg/L against Enterobacteriaceae, including most ESBL producers.1,2 Like all beta-lactam antibiotics, the time above MIC for free drug concentrations (ƒT>MIC) is the important PK-PD parameter correlating with its efficacy.11 When the beta-lactam antibiotic concentrations do not exceed the MIC for 40% to 50% of the dosing interval, the efficacy of a beta-lactam antibiotic can be compromised. When a cut-off of a ƒT>MIC of 40% is used, a Monte-Carlo simulation of the available data defines a clinical PK/PD breakpoint of 8 to 16 mg/L for temocillin.11-13 The available temocillin pharmacokinetics data (distribution, metabolism, and elimination) comes from studies performed in adults. It is mainly excreted unchanged (80%) in the urine by glomerular filtration and tubular secretion.3

Little is known about dosing and elimination of temocillin in children. The summary of product characteristics of temocillin proposes a daily dose of 25 - 50 mg/kg for paediatric use,14 but there are no studies that back-up this recommendation. This dose probably arises from scaling-down the typical adult daily dose of 2-4 g assuming an adult weight of 70kg. In the literature, the use of temocillin in paediatrics refers mainly to its clinical efficacy in the treatment of urinary tract infections.15,16 In the present hospital, temocillin is also used for the treatment of suspicion of cholangitis in cirrhotic paediatric patients, and as antibiotic prophylaxis following an hepatic transplant in children (both off-label indications). There is, therefore, a pressing need to explore the pharmacokinetics and pharmacodynamics of temocillin in the paediatric population, in order to provide clear guidance on an appropriate dosing regimen.

2. Study Objectives

1. Characterisation of the pharmacokinetics (PK) of temocillin (total and free concentrations) in 3 paediatric populations:

   1. children requiring antibiotic treatment for urinary tract infections
   2. cirrhotic children requiring antibiotic treatment due to suspicion of cholangitis
   3. children requiring antibiotic prophylaxis following an hepatic transplant
2. Proposal and development of a dosing schedule that can ensure therapeutic concentrations (40% ƒT > MIC) and optimize treatment chances of success.
3. Characterization of MICs of microbiological strains (when available) to temocillin.

3. Criteria for patients' selection 3.1 Inclusion Criteria

1. Male or female patient requiring temocillin

1. for the treatment of urinary tract infections, or
2. for the treatment of suspicion of cholangitis associated with cirrhosis, or
3. as antibiotic prophylaxis following an hepatic transplant. 2. Requirement of hospitalization (not for social or other non-medical reasons) for at least up to 5 days 3. Patients aged 6 months - 3 years at the beginning of the treatment with temocillin 4. Parents or legal representatives able to give written informed consent in accordance with GCP and local regulatory requirements, prior to any study procedure

   3.2 Exclusion Criteria
   1. Ig-E mediated allergy to penicillins
   2. Previous treatment with temocillin for the current cholangitis episode
   3. Diagnosis of Alagille syndrome
   4. Estimated life-expectance of < 5 days due to major co-morbid conditions
   5. Other serious illnesses, e.g. HIV, serious infections requiring other antibiotics, malignancy
   6. Patients with acute or chronic renal failure (eGFR < 30ml/min)
   7. Patients having participated in another study < 30 days before inclusion in the present study

   4. Investigational Plan 4.1 Study design and plan This is a prospective, open, non-interventional and monocentric study that will take place at the "Service de Gastro-entérologie pédiatrique" of the "Cliniques Universitaires St-Luc" in Brussels, Belgium. All patients eligible for treatment with temocillin will be evaluated and considered for inclusion in the study.

   For each of the 3 paediatric populations, a total of 30-35 patients eligible for participation will be included in the study. According to the manufacturer's information14 a dose of 25mg/kg (in cases of prophylaxis) or 50mg/kg (in cases of treatment) per day divided in 2 administrations will be used and administered by IV route. Blood samples will be drawn on day 1 and day 4 of treatment at 0.5, 2, 4, 8, 12 hours after dose administration. The patient's physician will decide on the duration of temocillin use.

   The expected total duration of the trial is 1 year (or more if patient enrollment is slow; number of patients to be included: 10-15 for each of the 3 paediatric populations; see next sentence for a justification of the addition of 15-20 patients per group after acceptance of an amendment to the initial protocol).

   An interim analysis on the first 14 patients from populations b and c suggested that the dose was too low to reach the pharmacodynamic target. An amendment has been submitted to the ethical committee of the cliniques universitaires Saint Luc and accepted (on 26/08/2019), to administer 25 mg/kg every 8 hours. This scheme will be used for the new patients to be recruted. 15-20 patients will be included with this new dosing regimen.

   4.2 Study procedures All blood samples (3mL each) will be taken from an arterial or venous catheter and collected in additive-free blood tubes. After blood clotting, they will be centrifuged and the serum will be frozen (-80°C) until analysis. Total concentration and free concentration will be determined by a validated High Pressure Liquid chromatography-Ultra Violet detection (HPLC-UV) method.12,17

   In addition, the following parameters will be recorded during study period: time of temocillin administration, patient's weight, renal and liver function markers (including total serum protein), infection markers, concomitant medications.

   5. Statistics

   The temocillin concentrations versus time data in serum will be analysed using a non-linear mixed effects modeling approach using a Nonlinear Mixed-Effects Modelling software (NONMEM version 7.3; ICON Development Solutions, Ellicott City, MD). The population pharmacokinetic model will then be defined, and used to simulated different dosing regimens with Monte Carlo simulations, that will be used for calculating the probability of target attainment (40% ƒT>MIC) for free concentration by MIC. Statistical significance is defined as P value of < 0.05. JMP version 11 software (SAS Institute, Cary, NC, USA) will be used for statistical analysis. If the clinical isolates for each patient are not available, the MIC distributions of the hospital will be considered for data analysis.

   6. Administrative Matters The trial will be carried out in compliance with the protocol, the principles laid down in the Declaration of Helsinki, in accordance with the International Committee on Harmonisation (ICH) Harmonised Tripartite Guideline for Good Clinical Practice (GCP) and in accordance with applicable regulatory requirements.

   6.1 Institutional Review Board / Independent Ethics Committee The trial will not be initiated before the protocol and informed consent and subject information form have been reviewed and received approval / favourable opinion from the local Institutional Review Board (IRB) or an Independent Ethics Committee (IEC).

   6.2 Informed Consent and Subject Information Prior to subject participation in the trial, written informed consent will be obtained from each subject's legally accepted representative according to the regulatory and legal requirements. Each signature must be dated by each signatory and the informed consent and any additional subject information form retained by the investigator as part of the study records. A signed copy of the informed consent and any additional subject information must be given to the subject's legally authorised representative.

   7. Timeframe: Outcome measure will be assessed within a maximum of 18 months.

ELIGIBILITY:
Inclusion Criteria:

* patient requiring temocillin

  1. for the treatment of urinary tract infections, or
  2. for the treatment of suspicion of cholangitis associated with cirrhosis, or
  3. as antibiotic prophylaxis following an hepatic transplant.
* patient requiring hospitalization (not for social or other non-medical reasons) for at least up to 5 days
* Parents or legal representatives able to give written informed consent in accordance with GCP and local regulatory requirements, prior to any study procedure

Exclusion Criteria:

1. Ig-E mediated allergy to penicillins
2. Previous treatment with temocillin for the current cholangitis episode
3. Diagnosis of Alagille syndrome
4. Estimated life-expectance of < 5 days due to major co-morbid conditions
5. Other serious illnesses, e.g. HIV, serious infections requiring other antibiotics, malignancy
6. Patients with acute or chronic renal failure (eGFR < 30ml/min)
7. Patients having participated in another study < 30 days before inclusion in the present study

Ages: 6 Months to 3 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 45 (Estimated)
Dates: Start 2016-02-17 (Actual); Primary Completion 2022-12-31 (Estimated); Study Completion 2022-12-31 (Estimated)

PRIMARY OUTCOMES:
Serum levels of temocillin | 18 months
  Characterisation of the pharmacokinetics (PK) of temocillin (total and free concentrations) in the 3 paediatric populations included

CONTACTS AND LOCATIONS:
Overall Officials: Françoise Van Bambeke, PharmD, PhD, Study Director — Université Catholique de Louvain
Locations (1):
- Cliniques universitaires St-Luc, Brussels, Belgium

REFERENCES:
- [Background] De Jongh R, Hens R, Basma V, Mouton JW, Tulkens PM, Carryn S. Continuous versus intermittent infusion of temocillin, a directed spectrum penicillin for intensive care patients with nosocomial pneumonia: stability, compatibility, population pharmacokinetic studies and breakpoint selection. J Antimicrob Chemother. 2008 Feb;61(2):382-8. doi: 10.1093/jac/dkm467. Epub 2007 Dec 10. PMID 18070831
- [Background] Livermore DM, Tulkens PM. Temocillin revived. J Antimicrob Chemother. 2009 Feb;63(2):243-5. doi: 10.1093/jac/dkn511. Epub 2008 Dec 18. PMID 19095679
- [Background] Miranda Bastos AC, Vandecasteele SJ, Tulkens PM, Spinewine A, Van Bambeke F. Development and validation of a high performance liquid chromatography assay for the determination of temocillin in serum of haemodialysis patients. J Pharm Biomed Anal. 2014 Mar;90:192-7. doi: 10.1016/j.jpba.2013.12.002. Epub 2013 Dec 12. PMID 24389461
- See also: Official Belgian "Summary of Product Characteristics" of temocillin (enter NEGABAN [trade name of temocillin] in the search window) — http://bijsluiters.fagg-afmps.be/?localeValue=en